CLINICAL TRIAL: NCT02853669
Title: Adductor Canal Block Versus Lumbar Plexus Block for Post Operative Pain Management After Total Knee Replacement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hassan Mohamed Ali, lecturer in anesthesia department Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: adductor canal
Record Dates: First submitted 2016-07-24; First posted 2016-08-03 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-07

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group (A) lumber plexus block (Experimental): Ultrasound-guided Lumber plexus Block (30 cc of 0.25% of bupivacaine, via a 22-gauge 2-inch Stimuplex A needle) with nerve stimulator confirmation.
  Interventions: Procedure: Ultrasound-guided Lumber Plexus Block
- Group (B) adductor canal block (Experimental): ultrasound-guided Adductor Canal Block (15 cc of 0.5% of bupivacaine)
  Interventions: Procedure: adductor canal block

INTERVENTIONS:
Procedure: Ultrasound-guided Lumber Plexus Block — (30 cc of 0.25% of bupivacaine, via a 22-gauge 2-inch Stimuplex A needle) with nerve stimulator confirmation. The type of motor response (e.g., quadriceps, patellar) and the minimum current needed were recorded. Ultrasound pictures (preinjection and postinjection) were obtained to verify proper local anesthetic placement.
  Arms: group (A) lumber plexus block
Procedure: adductor canal block — ultrasound-guided Adductor Canal Block (15 cc of 0.5% of bupivacaine)
  Other Names: saphenous nerve block
  Arms: Group (B) adductor canal block

SUMMARY:
Adductor canal block (ACB), Saphenous nerve block, which is a block of a purely sensory nerve which shares in nerve supply of knee joint has a hypothetical advantage of better pain management with less motor affection. Also, it has a clear anatomical landmark that will increase the success rate (femoral artery) (*).On the other hand, being a branch of the femoral nerve and far distal from the plexus, this can decrease the blocking effectiveness. Likewise, the great variation of the knee nerve supply.

This prospective double-blinded randomized controlled trial is comparing ultrasound guided adductor canal block (ACB) versus ultrasound-guided lumbar plexus block (LPB) in patients undergoing total knee arthroplasty aiming at decreasing post-operative pain, helping in early mobilization and better physiotherapy.

This study hypothesizes that ACB, compared with LPB, will exhibit less motor, weakness, fewer opioids consumption with the same or better pain score.

DETAILED DESCRIPTION:
This prospective double-blinded randomized controlled trial is comparing ultrasound guided adductor canal block (ACB) versus ultrasound-guided lumbar plexus block (LPB) in patients undergoing total knee arthroplasty aiming at decreasing post-operative pain, helping in early mobilization and better physiotherapy.

This study hypothesizes that ACB, compared with LPB, will exhibit less motor, weakness, fewer opioids consumption with the same or better pain score.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Age more than 25 and less than 80 were included

Exclusion Criteria:

* Patients with known allergy to the medications to be given
* ASA III, IV
* Age less than 25 or more than 80
* Dementia
* Deafness
* Psychological disease
* Difficult to communicate
* Cannot lay flat
* INR more than 1.5
* Low platelets (less than 100000/ml3) or with significant coagulopathy

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
pain | 2 hours
  pain assessment using visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Ali, LECTURER, Study Director — Anesthesia department, faculty of medicine ,Cairo university
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt